CLINICAL TRIAL: NCT01340547
Title: A Phase I Multicenter, Open-label Study of the Effect on QTc, Pharmacokinetics, Safety, and Preliminary Efficacy of Single-agent Palifosfamide-tris in Subjects With Advanced Solid Tumors
Brief Title: Effect on QTc, Pharmacokinetics, Safety, and Preliminary Efficacy of Single-agent Palifosfamide-tris in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM1005
Record Dates: First submitted 2011-04-13; First posted 2011-04-22 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Solid Tumors
Keywords: Phase I; Safety; PK; ECG QTc; Efficacy; Palifosfamide-tris; non-randomized
MeSH Terms: interventions — isophosphamide mustard; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single Arm, non-blinded, non-randomized
  Interventions: Drug: palifosfamide-tris; Drug: Normal Saline

INTERVENTIONS:
Drug: palifosfamide-tris — palifosfamide-tris IV infusion of 150 mg/m2 on Days 1, 2 and 3 every three weeks (21 day cycle)
  Other Names: isophosphoramide mustard-tris; Zymafos (TM)
Drug: Normal Saline — 0.9% Normal Saline 250 ml IV infusion on Cycle 1 Day -1

SUMMARY:
This is an open-label study of palifosfamide-tris administered intravenously on Days 1, 2, and 3 of a 21-day cycle to subjects with advanced solid tumors. Enrolled subjects will receive a placebo-control infusion on Day -1 and then commence palifosfamide-tris study treatment 24 hours later on Day 1.

Time-matched, intensive ECG monitoring will occur during and following placebo and palifosfamide-tris infusions on Days -1, 1, 2, 3 and 8. Generation of ECG data for study analysis will be performed in a blinded fashion at a central ECG laboratory.

Blood and urine sampling to characterize the pharmacokinetics of palifosfamide-tris will be performed on Days 1 through 8 of Cycle 1.

ELIGIBILITY:
Inclusion criteria:

1. Male or female subjects, age ≥ 18 years, who have provided written informed consent prior to completing any study specific procedure.
2. Histologically or cytologically confirmed solid tumor that has progressed following available standard therapies or for which no standard therapy exist.
3. Measurable or non-measurable disease by RECIST version 1.1
4. Must have recovered from toxic effects of prior cancer treatment to ≤ Grade1per CTCAE v4.0, with the exception of any alopecia.
5. ECOG Performance Status of 0 or 1.
6. Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements:

   1. Hemoglobin ≥9.0 g/dL.
   2. Absolute neutrophil count (ANC) ≥1,500/uL.
   3. Platelet count ≥100,000/uL.
   4. Total bilirubin ≤1.5 x upper limit of normal (ULN)
   5. ALT and AST ≤2.5 x ULN. For subjects with documented liver metastases, ALT and AST ≤5×ULN.
   6. International Normalized Ratio (INR) and activated partial thromboplastin time [PTT] <1.5 x ULN, if not therapeutically anticoagulated. Subjects who are being therapeutically anticoagulated with an agent such as Coumadin (warfarin sodium) or subcutaneous heparin may be included provided there is no prior evidence of underlying abnormality in coagulation parameters, screening test results are in appropriate therapeutic range, and anticoagulation regimen is stable and closely monitored.
   7. Estimated glomerular filtration rate (eGRF) ≥60 mL/minute/1.73 m2.
7. Male and female subjects must agree to use a highly reliable method of birth control (expected failure rate less than 5% per year) from the screening visit through 28 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects who have received prior chemotherapy, radiation therapy or any investigational agent within 28 days prior to the first dose of study drug.
2. Unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a subject and/or their compliance with the protocol. Examples include, but are not limited to, unstable angina, congestive heart failure, recent (within 2 months of screening) myocardial infarction, ongoing maintenance therapy for life-threatening ventricular arrhythmia, uncontrolled asthma, HIV/AIDS without adequate anti-viral therapy, evidence of hepatic pathology due to or consistent with infection with a chronic hepatitis virus, uncontrolled major seizure disorder, or electrolyte imbalances.
3. Presence of, or history of any illness or injury to the urinary tract (renal or post-renal) which may make the subject more susceptible to acute renal insufficiency in the case of potential renal adverse events. Types of injury or illness might include a history of polycystic renal disease, nephrectomy, renal transplant, acute or chronic renal failure.
4. Active infection requiring systemic antibacterial, antifungal, or antiviral therapy within 2 weeks of the first dose of study drug. Subjects with HIV who are on effective anti-viral therapy or subjects with chronic herpes infections who use intermittent suppressive antiviral therapy for viral outbreaks may be included.
5. Major surgery within 4 weeks prior to start of treatment.
6. Documented symptomatic brain metastases. Screening for brain lesions by CT or MRI is not required for potential subjects; however, if there are any neurological signs or symptoms consistent with brain metastases, then a brain CT or MRI should be performed as clinically indicated.
7. Currently pregnant or nursing.
8. Subjects with implantable pacemaker or automatic implantable cardioverter defibrillator.
9. Conditions that make the screening ECG repolarization difficult to interpret, or showing significant abnormalities. This includes, but is not limited to: high degree AV block, pace-maker, atrial fibrillation or flutter, prolonged QTc >500ms on repeat measurements (e.g., 2 out of 3 ECGs), or bradycardia (defined as ≤ 50 beats/minute).
10. Subjects who will be receiving medications that prolong the QT interval with a risk of causing Torsades de Pointes during the time period beginning 1 week prior to and during the Intensive ECG monitoring period (i.e., Cycle 1, Day -8 through Day 8).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
ECG QTc intervals of patients who receive palifosfamide-tris | Cycle 1 Days -1,1, 2, 3,8
  To assess the effect of single-agent palifosfamide-tris on QTc intervals.
Blood sampling to characterize the pharmacokinetics of palifosfamide-tris | Cycle 1, Day 1, 2, 3, 4, 8
  To assess the pharmacokinetic profile of single-agent palifosfamide-tris.

SECONDARY OUTCOMES:
Safety and tolerability of palifosfamide-tris measured in amount, type, severity and relatedness of Adverse Events | Duration of time patient is on study, expected average of 5 months
  To assess the safety and tolerability of single-agent palifosfamide-tris.
Preliminary efficacy of palifosfamide-tris as it pertains to cancer tumor growth | Duration of time patient is on study, expected average of 5 months
  To obtain preliminary efficacy data as defined by objective response rate (ORR); progression-free survival (PFS); and durability of response in subjects with advanced solid tumors when treated with single-agent palifosfamide-tris.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas